CLINICAL TRIAL: NCT02994043
Title: Dismantling MBRP: Identifying Critical Neuroimmune Mechanisms of Action.
Brief Title: Alcohol, Inflammation, and Mindfulness Study (AIM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2550; R01AA024632 (NIH)
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRP (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Relapse Prevention Therapy
- RP (Active Comparator)
  Interventions: Behavioral: Relapse Prevention Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Relapse Prevention Therapy — An 8-week, outpatient psychotherapy that combines mindfulness components with relapse prevention.
  Arms: MBRP
Behavioral: Relapse Prevention Therapy — An 8-week, outpatient psychotherapy that uses cognitive-behavioral components to reduce alcohol-related consequences.
  Arms: RP

SUMMARY:
The goal of the AIM Study is to examine the effectiveness of Mindfulness Based Relapse Prevention (MBRP) versus Relapse Prevention (RP) for the treatment of Alcohol Use Disorders (AUD) by implementing an 8-week long intervention and examining neurobiological, immunological, and epigenetic characteristics of AUD.

DETAILED DESCRIPTION:
This study was designed to evaluate the effect of two outpatient, individually-administered, psychosocial interventions (Relapse Prevention vs. Mindfulness-Based Relapse Prevention). Participants are recruited via mass media advertisements, flyers, and local outreach to clinical providers that do not address substance use. We will recruit 226 individuals. Our previous experience with clinical trials, as well as the experience of our research team members with these interventions support the feasibility of recruiting approximately 50 patients per year. This sample size provides adequate statistical power for the research questions undertaken.

Participants are screened over the telephone and invited into the laboratory for a baseline assessment. Immediately after the baseline assessment, they are randomized to a therapist and then to a treatment condition. At the end of each year, the distribution of participants across conditions and therapists are evaluated for imbalances. If attrition has resulted in an imbalance across conditions, the randomization procedure will be adjusted to ensure equal numbers of participants in RP and MBRP.

Within a week of completing the baseline assessments, participants are seen by their individual therapist for a motivational interviewing, goal-setting session. After the goal-setting session, the eight-session MBRP or RP treatments are administered. To ensure that therapists adhere to treatment manuals, a checklist is provided consisting of the primary content addressed each session (four to seven primary content pieces each session). Further, questionnaires assessing mindfulness practice and facets of mindfulness (e.g., being nonjudgmental, nonreactive) are administered at each assessment. At the most recent RPPR, these questionnaires validated that participants in the MBRP condition were increasing in some facets of mindfulness during treatment (and up to three months after treatment).

We estimate that the completion of assessments and procedures across the duration of the trial, excluding therapy sessions, will total about 15 hours of time. To compensate subjects for their time and travel costs, each subject will be paid $300 if they complete all sessions.

We will conduct extensive analyses of any attrition encountered in the project to determine bias. However, note that in each of the analyses described herein, we will have the capability of using modern approaches to the handling of missing data including full information maximum likelihood estimation of missing data within Proc Mixed in SAS and within EQS.

The distributional properties of all continuously scaled variables will be examined for skewness and kurtosis to determine the need for normalizing transformations or for alternations to our analysis plan (i.e., generalized estimating equations or robust estimation) prior to the primary analyses.

To confirm the validity of random assignment, pretest equivalence of the two treatment conditions across demographics, drinking history, smoking, and all other baseline measures will be assessed via t-tests on continuous items and c2 tests of categorical items. We will use the Bonferroni approach to correct for alpha inflation with a familywise alpha of .05. Any variables on which the two groups are unequal at pretest will be covariates in all further analyses.

Attrition analyses will be conducted after each follow-up data collection effort to provide assurance that differential attrition by treatment condition has not occurred. Following previously published procedures, a series of ANOVAs of treatment (MBRP versus RP) X retention (retained, not retained) will be conducted on continuous baseline measures. Significant treatment X retention interactions identify measured variables on which differential attrition may have occurred. The logit model analog procedure will be applied to categorical baseline measures to test for differential attrition on categorical variables such as gender and ethnicity. We will conduct these analyses to assure that differential attrition by treatment condition does not account for any of the effects of the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Have a primary Diagnostic Statistical Manual-V (DSM-V) diagnosis of alcohol use disorder;
2. Must be within 10 days of last drink;
3. Must have been drinking heavily (criteria dependent upon individual?s age, gender, and BMI) for a consistent period of time;
4. Must have a breath alcohol level of 0 at screening;
5. Must have a Clinical Institute Withdrawal Assessment (CIWA) score less than 8 (indicating no need for medical detox);
6. Must have expressed a desire during their initial screen to reduce the number of drinks they regularly consume

Exclusion Criteria:

1. Currently taking any medications for the treatment of psychiatric disorders, including substance use disorders, mood disorders, and psychosis;
2. Pregnant, as indicated by a pregnancy test which will be administered at baseline;
3. Positive for, sedatives, opiates, cocaine, or amphetamine on drug screen at baseline;
4. Meets criteria for psychotic disorder, bipolar disorder, or a major depressive episode

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Hutchison, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skrzynski CJ, Karoly H, Ellingson JM, Hagerty SL, Bryan AD, Hutchison KE. Comparing the Efficacy of Mindfulness-Based Relapse Prevention Versus Relapse Prevention for Alcohol Use Disorder: A Randomized Control Trial. J Stud Alcohol Drugs. 2023 Jul;84(4):560-569. doi: 10.15288/jsad.21-00392. Epub 2023 Feb 1. PMID 36971735
- [Derived] Karoly HC, Skrzynski CJ, Moe EN, Bryan AD, Hutchison KE. Exploring relationships between alcohol consumption, inflammation, and brain structure in a heavy drinking sample. Alcohol Clin Exp Res. 2021 Nov;45(11):2256-2270. doi: 10.1111/acer.14712. Epub 2021 Sep 22. PMID 34523725
- [Derived] Karoly HC, Ross JM, Prince MA, Zabelski AE, Hutchison KE. Effects of cannabis use on alcohol consumption in a sample of treatment-engaged heavy drinkers in Colorado. Addiction. 2021 Sep;116(9):2529-2537. doi: 10.1111/add.15407. Epub 2021 Jan 26. PMID 33464670

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness-Based Relapse Prevention: Mindfulness-Based Relapse Prevention Therapy: An 8-week, outpatient psychotherapy that uses cognitive-behavioral components to reduce alcohol-related consequences.
- Relapse Prevention: Relapse Prevention Therapy: An 8-week, outpatient psychotherapy that combines mindfulness components with relapse prevention.
Period: Overall Study
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Started | 90 | 92
Completed | 71 | 75
Not Completed | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- MBRP: Mindfulness Plus Relapse Prevention Therapy: An 8-week, outpatient psychotherapy that uses cognitive-behavioral components to reduce alcohol-related consequences.
- Total: Total of all reporting groups
Arm/Group | MBRP | Relapse Prevention | Total
Number analyzed (Participants) | 90 | 92 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.0) | 44.2 (10.3) | 44.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 50 | 44 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 84 | 84 | 168
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days at Baseline
Description: Timeline Follow-back (TLFB) measure of heavy drinking days in the last month (4+ for women, 5+ for men)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Heavy Drinking Days
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Number analyzed (Participants) | 90 | 92
Heavy Drinking Days | 12.6 (10.3) | 11.7 (10.5)

2. Primary Outcome: Heavy Drinking Days at Week 4
Description: Timeline Follow-back (TLFB) measure of heavy drinking days in the last month (4+ for women, 5+ for men)
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Heavy Drinking Days
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Number analyzed (Participants) | 80 | 87
Heavy Drinking Days | 7.8 (8.2) | 7.6 (8.5)

3. Primary Outcome: Heavy Drinking Days at Week 8
Description: Timeline Follow-back (TLFB) measure of heavy drinking days in the last month (4+ for women, 5+ for men)
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: Heavy Drinking Days
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Number analyzed (Participants) | 71 | 75
Heavy Drinking Days | 6.5 (7.9) | 5.3 (7.6)

4. Primary Outcome: Heavy Drinking Days at Week 20
Description: Timeline Follow-back (TLFB) measure of heavy drinking days in the last month (4+ for women, 5+ for men)
Time Frame: Week 20
Measure: Mean (Standard Deviation); unit: Heavy Drinking Days
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Number analyzed (Participants) | 61 | 57
Heavy Drinking Days | 6.1 (8.0) | 7.3 (8.8)

5. Primary Outcome: Heavy Drinking Days at Week 32
Description: Timeline Follow-back (TLFB) measure of heavy drinking days in the last month (4+ for women, 5+ for men)
Time Frame: Week 32
Measure: Mean (Standard Deviation); unit: Heavy Drinking Days
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
Number analyzed (Participants) | 58 | 50
Heavy Drinking Days | 4.7 (6.5) | 7.7 (8.2)

ADVERSE EVENTS:
Time Frame: 32 Weeks
Arm/Group | Mindfulness-Based Relapse Prevention | Relapse Prevention
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/92
Other Adverse Events (participants affected / at risk) | 0/90 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02994043/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT02994043/ICF_001.pdf